CLINICAL TRIAL: NCT04890964
Title: Mapping the Impact of the Montage of the Transcranial Direct Current Stimulation at Home at Cortical and Psycho-cognitive Functions, Functional Capacity and Biological Rhythm in the Fibromyalgia: A Randomized, Factorial, Clinical Trial
Brief Title: Montage of HTDCS in Psycho-cognitive Functions in FM
Acronym: HFTDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36995020.3.0000.5327
Record Dates: First submitted 2021-02-24; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; chronic pain; tDCS; TMS; BDNF; cortical connectivity
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: HB-a-tDCS - M1 (n=33); HB-s-tDCS - M1 (n=17); HB-a-tDCS-DLPFC (n=33); HB-a-tDCS- DLPFC (n=17)
Who Masked: Participant, Care Provider, Investigator
Masking Description: A randomized, double-blind, factorial, parallel-group, controlled trial with simulated treatment will be performed. The study follows the CONSORT guideline and will be registered in the ClinicalTrials.gov database: Home
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcranial Direct Current Stimulation (tDCS), Active Stimulation - DLPFC (Active Comparator): Participants received Active stimulation 20 minutes daily for 20 days, and 4 times after continuous stimulation, every 15 days.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Transcranial Direct Current Stimulation (tDCS), Sham Stimulation - DLPFC (Sham Comparator): Participants received Sham stimulation 20 minutes daily for 20 days, and 4 times after continuous stimulation, every 15 days.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Transcranial Direct Current Stimulation (tDCS), Active Stimulation - M1 (Active Comparator): Participants received Active stimulation 20 minutes daily for 20 days, and 4 times after continuous stimulation, every 15 days.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Transcranial Direct Current Stimulation (tDCS), Sham Stimulation - M1 (Placebo Comparator): Participants received Sham stimulation 20 minutes daily for 20 days, and 4 times after continuous stimulation, every 15 days.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — A stimulation device, that releases 2.0mA current by a 35 cm2 electrode direct located on a specific location on the scalp for 20 minutes
  Other Names: tDCS; Non Invasive Brain Stimulation (NIBS)

SUMMARY:
This study aims to map the impact of anodic transcranial direct current stimulation (tDCS) for prolonged home use applied to the primary motor cortex and the left dorsolateral prefrontal córtex (DLPFC), compared to the respective treatments simulated in fibromyalgia.

DETAILED DESCRIPTION:
This study aims to map the impact of anodic tDCS for prolonged home use applied to the primary motor cortex and the left dorsolateral prefrontal córtex (DLPFC), compared to the respective treatments simulated in fibromyalgia, targeting the outcomes of the following axes: (1) pain intensity and functional capacity; (2) psycho cognitive functions; (3) neurophysiological markers; (4) biological rhythm markers; (5) to map the potential of neurophysiological markers, biological rhythm and history of trauma in childhood and adolescence in functional capacity, depressive symptoms and working memory tests.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 65 years; who can read and write, with a confirmed diagnosis of FM according to the criteria of the American College of Rheumatology (2010-2016). Pain score equal to or greater than six on the Numeric Pain Scale (NPS 0-10) on most days in the last 3 months.

Exclusion Criteria:

* Living outside Porto Alegre area and pregnancy.
* Contraindications to TMS and tDCS: metallic implant in the brain; medical devices implanted in the brain, cardiac pacemaker; aneurysmal clip; metallic cochlear prosthesis, ear implants, and non-removable hearing aids; infusion pumps (including implantable); cranial halos. Pregnant women, shift work, use of exogenous melatonin, history of alcohol or drug abuse in the last 6 months, neurological pathologies, history of head trauma or neurosurgery, decompensated systemic chronic diseases, chronic inflammatory diseases (lupus, rheumatoid arthritis, Reiter's syndrome), personal history of cancer, past or under treatment.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We have chosen women over men, due to the prevalence of the disease that we are researching and also because the symptoms characteristics are more homogeneous.
Enrollment: 66 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
level of pain | Up to 60 minutes before and after tDCS stimulation
  response on the Numeric Verbal Scale (NPS) from 0-10 during the conditioning stimulus

SECONDARY OUTCOMES:
Psychocognitive functions | Pre and Pos 20 days Intervention
  episodic memory measured by Rey Verbal test
circadian rhythmicity | Pre and Pos 20 days Intervention
  urinary 6-sulfatoxymelatonin levels
Effect of tDCS over DLPFC on cognitive function. | Pre and Pos 20 days Intervention
  Cortical connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, Dr, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil